CLINICAL TRIAL: NCT03426111
Title: Multicenter, Randomized, Controlled and Double-blind Study of Efficacy and Safety of Endoscopic Gastric Tubulization in Patients With Non-alcoholic Steatohepatitis (NASH-APOLLO).
Acronym: NASH-APOLLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Jose Luis Calleja, Professor and Head of Hepatology Unit of Puerta de Hierro University Hospital, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI17-00499
Record Dates: First submitted 2018-01-09; First posted 2018-02-08 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
Keywords: Non-Alcoholic Fatty Liver Disease; NASH; Obesity; Endoscopic gastric tubulization; Non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized,controlled and double-blind study with two parallel arms, placebo (normal endoscopy and lifestyle modification) or endoscopic gastric tubulization with OverStitch® system (Apollo Endosurgery, Austin, TX, USA) and lifestyle modification.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Diagnostic upper endoscopy plus lifestyle modification.
  Interventions: Behavioral: Lifestyle modification
- Treatment (Active Comparator): Endoscopic gastric tubulization with OverStitch® system (Apollo Endosurgery, Austin, TX, USA) plus lifestyle modification.
  Interventions: Device: Endoscopic Gastric Tubulization with OverStitch® system (Apollo Endosurgery, Austin, TX, USA); Behavioral: Lifestyle modification

INTERVENTIONS:
Device: Endoscopic Gastric Tubulization with OverStitch® system (Apollo Endosurgery, Austin, TX, USA) — This endoscopic technique is defined as a gastric restriction by means of sutures of the entire gastric wall, transmurally, in order to simulate a gastric sleeve, in the same way as sleeve gastrectomy surgery. Gastroplasty is performed using an endoscopic suture system (OverStitch, Apollo Endosurgery Inc., Austin, Texas, USA) inserted into a dual-channel endoscope (GIF-2T160, Olympus Medical Systems Corp., Tokyo, Japan).
  Arms: Treatment
Behavioral: Lifestyle modification — Hypocaloric diet and moderate physical exercise

SUMMARY:
Nonalcoholic steatohepatitis is a growing public health problem affecting over 5% of the population. These patients are at increased risk of cardiovascular and liver-related death and have higher rates of malignancy.

The currently standard of care is weight loss and physical exercise, with histological and analytical improvement in patients achieving a 5-10% reduction in body weight. However, less than 25% of the subjects achieve this goal. In obese patients , restrictive surgical treatments and gastric bypass have been successful in improving the metabolic syndrome, insulin resistance and liver histology.

Currently, less invasive and less costly endoscopic techniques are being developed. These techniques also achieve a gastric restriction with similar results than bariatric surgery. One of these is the OverStitch® system (Apollo Endosurgery, Austin, TX, USA). Our aim is to evaluate the efficacy and safety of this method in the improvement of liver histology in obese patients with nonalcoholic steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged between 18 and 75 years (inclusive) at the time of the first screening visit.
2. They must provide signed written informed consent and agree to comply the study protocol
3. Body mass index> 30 kg / m².
4. Histological confirmation of steatohepatitis in a diagnostic liver biopsy (biopsy obtained in the 6 months prior to randomization or during the selection period) with at least a score of 1 in each component of the NAS score (steatosis with a score of 0 to 3, degeneration by ballooning with a score of 0 to 2 and lobular inflammation with a score of 0 to 3) and fibrosis of 0 to <4, according to the staging system of CRN fibrosis on NASH.
5. NAS score ≥ 4.
6. For patients without fibrosis or with stage 1 fibrosis, the NAS score≥5 and one of the following conditions (metabolic syndrome (definition NCEP ATP III), DM type II, HOMA-IR> 6).
7. The liver biopsy should have been done with a 16 G trucut needle and the minimum size should be 25 mm.

Exclusion Criteria:

1. Known heart failure (Grade I to IV of the classification of the New York Heart Association).
2. History of effective bariatric surgery in the 5 years prior to selection.
3. Patients with a history of clinically significant acute cardiac event in the 6 months prior to selection, such as: acute cardiovascular event, cerebrovascular accident, transient ischemic attack, or coronary heart disease (angina pectoris, myocardial infarction, revascularization procedures).
4. Weight loss of more than 5% in the 6 months prior to randomization.
5. Liver cirrhosis.
6. Non-cirrhotic portal hypertension.
7. Recent or current background of significant consumption of alcoholic beverages (<5 years). In the case of men, significant consumption is usually defined as more than 30 g of pure alcohol per day. In the case of women, it is usually defined as more than 20 g of pure alcohol per day.
8. Esophagogastric varices.
9. Hepatocellular carcinoma
10. Portal thrombosis.
11. Pregnancy.
12. Refusal to give informed consent.
13. Any medical condition that could reduce life expectancy to less than 2 years, including known cancers.
14. Signs of any other unstable or clinically significant immunological, endocrine, hematological, gastrointestinal, neurological, neoplastic or psychiatric disease without treatment.
15. Instability or mental incompetence, so that the validity of the informed consent or the ability to comply with the study are uncertain.

    In addition to the above criteria, the patient must not present any of the following biological exclusion criteria:
16. Antibodies positive for the human immunodeficiency virus.
17. Aspartate aminotransferase (AST) and / or ALT> 10 x upper limit of normal (ULN).
18. Total bilirubin> 25 μmol / l (1.5 mg / dl).
19. Standardized international index> 1.4.
20. Platelet count <100 000 / mm3.
21. Serum creatinine levels> 135 μmol / l (> 1.53 mg / dl) in men and> 110 μmol / l (> 1.24 mg / dl) in women.
22. Significant renal disease, including nephritic syndrome, chronic kidney disease (patients with markers of hepatic injury or estimated glomerular filtration rate [eGFR] of less than 60 ml / min / 1.73 m2). If an abnormal value is obtained at the first screening visit, the eGFR measurement may be repeated before randomization within the following time frame: minimum 4 weeks after the initial test and maximum 2 weeks before the expected randomization. An abnormal repeated eGFR (less than 60 ml / min / 1.73 m2) leads to exclusion from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of gastric tubulization + modification in lifestyle for 72 weeks compared to standard treatment / placebo in the resolution of NASH without worsening of fibrosis. | 72 weeks
  NASH resolution is defined as the disappearance of ballooning and the disappearance or persistence of minimal lobular inflammation (grade 0 or 1) The worsening of fibrosis is defined as the progression of at least one stage.

SECONDARY OUTCOMES:
Number of patients with improvement of fibrosis according to the CRN score NASH. | 72 weeks
  to evaluate other histological changes after 72 weeks of treatment (CRN)
Non alcoholic fatty liver disease (NASH) activity score (NAS). | 72 weeks
  Number of patients with improvement in histological scores CRN score on NASH (NAS)
steatosis-activity-fibrosis index score (steatosis activity fibrosis, SAF). | 72 weeks
  Number of patients with improvement in the SAF score.
Cardiovascular and death events related to the liver | 72 weeks
  To evaluate the CV events in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo
Changes in liver enzymes | 72 weeks
  To evaluate liver enzymes in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo
Changes in the noninvasive markers of fibrosis and steatosis | 72 weeks
  To evaluate the noninvasive markers in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo
Changes in lipid parameters | 72 weeks
  To evaluate the lipid parameters in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo
Variation in body weight | 72 weeks
  To evaluate body weight in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo
Biomarkers of endothelial and macrophage dysfunction | 72 weeks
  To evaluate macrophage function in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo
Changes in markers of homeostasis of glucose and insulin resistance | 72 weeks
  To evaluate the glucose metabolism in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo
Changes in cardiovascular risk profile | 72 weeks
  To evaluate cardiovascular risk profile in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo
Changes in quality of life (abbreviated health questionnaire SF-36). | 72 weeks
  To evaluate the following endpoints in patients treated with gastric endoscopic tubulization + lifestyle modification with respect to lifestyle modification / placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Luis Calleja, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Wanless IR, Lentz JS. Fatty liver hepatitis (steatohepatitis) and obesity: an autopsy study with analysis of risk factors. Hepatology. 1990 Nov;12(5):1106-10. doi: 10.1002/hep.1840120505. PMID 2227807
- [Background] Stepanova M, Rafiq N, Makhlouf H, Agrawal R, Kaur I, Younoszai Z, McCullough A, Goodman Z, Younossi ZM. Predictors of all-cause mortality and liver-related mortality in patients with non-alcoholic fatty liver disease (NAFLD). Dig Dis Sci. 2013 Oct;58(10):3017-23. doi: 10.1007/s10620-013-2743-5. Epub 2013 Jun 18. PMID 23775317
- [Background] Michelotti GA, Machado MV, Diehl AM. NAFLD, NASH and liver cancer. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):656-65. doi: 10.1038/nrgastro.2013.183. Epub 2013 Oct 1. PMID 24080776
- [Background] Adams LA, Sanderson S, Lindor KD, Angulo P. The histological course of nonalcoholic fatty liver disease: a longitudinal study of 103 patients with sequential liver biopsies. J Hepatol. 2005 Jan;42(1):132-8. doi: 10.1016/j.jhep.2004.09.012. PMID 15629518
- [Background] Angulo P. Diagnosing steatohepatitis and predicting liver-related mortality in patients with NAFLD: two distinct concepts. Hepatology. 2011 Jun;53(6):1792-4. doi: 10.1002/hep.24403. No abstract available. PMID 21557278
- [Background] Neuschwander-Tetri BA. Non-alcoholic fatty liver disease. BMC Med. 2017 Feb 28;15(1):45. doi: 10.1186/s12916-017-0806-8. PMID 28241825
- [Background] Gallego-Duran R, Cerro-Salido P, Gomez-Gonzalez E, Pareja MJ, Ampuero J, Rico MC, Aznar R, Vilar-Gomez E, Bugianesi E, Crespo J, Gonzalez-Sanchez FJ, Aparcero R, Moreno I, Soto S, Arias-Loste MT, Abad J, Ranchal I, Andrade RJ, Calleja JL, Pastrana M, Iacono OL, Romero-Gomez M. Imaging biomarkers for steatohepatitis and fibrosis detection in non-alcoholic fatty liver disease. Sci Rep. 2016 Aug 12;6:31421. doi: 10.1038/srep31421. PMID 27514671
- [Background] Barr J, Caballeria J, Martinez-Arranz I, Dominguez-Diez A, Alonso C, Muntane J, Perez-Cormenzana M, Garcia-Monzon C, Mayo R, Martin-Duce A, Romero-Gomez M, Lo Iacono O, Tordjman J, Andrade RJ, Perez-Carreras M, Le Marchand-Brustel Y, Tran A, Fernandez-Escalante C, Arevalo E, Garcia-Unzueta M, Clement K, Crespo J, Gual P, Gomez-Fleitas M, Martinez-Chantar ML, Castro A, Lu SC, Vazquez-Chantada M, Mato JM. Obesity-dependent metabolic signatures associated with nonalcoholic fatty liver disease progression. J Proteome Res. 2012 Apr 6;11(4):2521-32. doi: 10.1021/pr201223p. Epub 2012 Mar 15. PMID 22364559
- [Background] Alkhouri N, Feldstein AE. Noninvasive diagnosis of nonalcoholic fatty liver disease: Are we there yet? Metabolism. 2016 Aug;65(8):1087-95. doi: 10.1016/j.metabol.2016.01.013. Epub 2016 Feb 2. PMID 26972222
- [Background] Nobili V, Parkes J, Bottazzo G, Marcellini M, Cross R, Newman D, Vizzutti F, Pinzani M, Rosenberg WM. Performance of ELF serum markers in predicting fibrosis stage in pediatric non-alcoholic fatty liver disease. Gastroenterology. 2009 Jan;136(1):160-7. doi: 10.1053/j.gastro.2008.09.013. Epub 2008 Sep 20. PMID 18992746
- [Background] Ratziu V, Massard J, Charlotte F, Messous D, Imbert-Bismut F, Bonyhay L, Tahiri M, Munteanu M, Thabut D, Cadranel JF, Le Bail B, de Ledinghen V, Poynard T; LIDO Study Group; CYTOL study group. Diagnostic value of biochemical markers (FibroTest-FibroSURE) for the prediction of liver fibrosis in patients with non-alcoholic fatty liver disease. BMC Gastroenterol. 2006 Feb 14;6:6. doi: 10.1186/1471-230X-6-6. PMID 16503961
- [Background] Vilar-Gomez E, Martinez-Perez Y, Calzadilla-Bertot L, Torres-Gonzalez A, Gra-Oramas B, Gonzalez-Fabian L, Friedman SL, Diago M, Romero-Gomez M. Weight Loss Through Lifestyle Modification Significantly Reduces Features of Nonalcoholic Steatohepatitis. Gastroenterology. 2015 Aug;149(2):367-78.e5; quiz e14-5. doi: 10.1053/j.gastro.2015.04.005. Epub 2015 Apr 10. PMID 25865049
- [Background] Klebanoff MJ, Corey KE, Chhatwal J, Kaplan LM, Chung RT, Hur C. Bariatric surgery for nonalcoholic steatohepatitis: A clinical and cost-effectiveness analysis. Hepatology. 2017 Apr;65(4):1156-1164. doi: 10.1002/hep.28958. Epub 2017 Feb 21. PMID 27880977
- [Background] Mummadi RR, Kasturi KS, Chennareddygari S, Sood GK. Effect of bariatric surgery on nonalcoholic fatty liver disease: systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2008 Dec;6(12):1396-402. doi: 10.1016/j.cgh.2008.08.012. Epub 2008 Aug 19. PMID 18986848
- [Background] ASGE Bariatric Endoscopy Task Force; ASGE Technology Committee; Abu Dayyeh BK, Edmundowicz SA, Jonnalagadda S, Kumar N, Larsen M, Sullivan S, Thompson CC, Banerjee S. Endoscopic bariatric therapies. Gastrointest Endosc. 2015 May;81(5):1073-86. doi: 10.1016/j.gie.2015.02.023. Epub 2015 Mar 28. No abstract available. PMID 25828245
- [Background] ASGE/ASMBS Task Force on Endoscopic Bariatric Therapy; Ginsberg GG, Chand B, Cote GA, Dallal RM, Edmundowicz SA, Nguyen NT, Pryor A, Thompson CC. A pathway to endoscopic bariatric therapies. Gastrointest Endosc. 2011 Nov;74(5):943-53. doi: 10.1016/j.gie.2011.08.053. No abstract available. PMID 22032311
- [Derived] Abad J, Llop E, Arias-Loste MT, Burgos-Santamaria D, Martinez Porras JL, Iruzubieta P, Graus J, Ruiz-Antoran B, Sanchez Yuste MR, Romero-Gomez M, Albillos A, Crespo J, Calleja JL. Endoscopic Sleeve Gastroplasty Plus Lifestyle Intervention in Patients With Metabolic Dysfunction-associated Steatohepatitis: A Multicenter, Sham-controlled, Randomized Trial. Clin Gastroenterol Hepatol. 2025 Aug;23(9):1556-1566.e3. doi: 10.1016/j.cgh.2024.10.027. Epub 2024 Dec 16. PMID 39694202